CLINICAL TRIAL: NCT03177473
Title: A Multi-Center, Open-Label, Prospective Study of CervicalStim Device™ as Adjunctive Care Following Cervical Fusion
Brief Title: Study Using the CervicalStim Device Following Cervical Fusion
Status: Completed | Type: Observational
Sponsor: Orthofix Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CP-1703CSPM
Record Dates: First submitted 2017-04-27; First posted 2017-06-06 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Vertebral Cervical Fusion Syndrome; Degenerative Disc Disease
Keywords: degenerative disc disease; CervicalStim devic; cervical; cervical fusion
MeSH Terms: conditions — Klippel-Feil Syndrome; Intervertebral Disc Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- CervicalStim PEMF group: all subjects will receive active CervicalStim bone growth stimulator
  Interventions: Device: CervicalStim bone growth stimulator

INTERVENTIONS:
Device: CervicalStim bone growth stimulator — Orthofix CervicalStim bone growth stimulator

SUMMARY:
This study examines the effect of adjunctive use of the CervicalStim bone growth stimulator on cervical fusion rate in high risk subjects who have undergone cervical fusion surgery. All participants will wear the bone growth stimulator every day for 4 hours/day for 6 months.

DETAILED DESCRIPTION:
The purpose of this post market prospective study is to examine the effect of the adjunctive use of the Orthofix CervicalStim device on cervical fusion rate in high risk subjects who have undergone cervical fusion surgery. High risk subjects are those who are having a multi-level (2 or more) cervical fusion, who are smokers, who are diabetic or those who are osteoporotic. Because this is a post market prospective study, subjects who are enrolled in this study will be identified by the Investigator as needing cervical fusion surgery and asked to participate in a study looking at the efficacy of cervical fusion with adjunctive use of the CervicalStim bone growth simulator. The type of cervical fusion surgery performed is up to the Investigator; the subjects in the study must be agreeable to using the bone growth stimulator for 6 months post-surgery. The subjects will be followed for 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, ≥ 18 years of age at the time of Informed Consent.
2. Requires a cervical fusion surgery within 30 days of Informed Consent signing.

   a. Surgical approach is at the physician's discretion.
3. Subject has one or more high risk factors:

   1. Is currently using nicotine
   2. multi-level cervical fusion surgery planned
   3. Prior failed fusion at any cervical level
   4. Subject reported diabetes
   5. Subject reported osteoporosis
4. Body mass index ≤ 45 kg/m2 at the time of consent.
5. Must have reliable access to an iPhone or an iPad with Wi-Fi access for downloading the free device-specific app (iPhone 5S or higher, iPad, iPad Pro, iPad mini or iTouch using iOS v.9.3 or later).

   a. When the android version of the mobile app for the CervicalStim device becomes available (estimated to be Dec. 2017), subjects who have reliable access to devices using android operating systems will be eligible for study inclusion.
6. Able and willing to complete electronic questionnaires and able to read and understand study instructions in English.
7. Able and willing to comply with the study plan and able to understand and sign the study-specific Informed Consent Form (ICF).

Exclusion Criteria:

1. Current alcoholism and/or any known current addiction to pain medications.
2. Any active malignancy or prior history of malignancy within last 5 years prior to fusion (except basal cell carcinoma of the skin).
3. Any clinically significant finding that places the subject at health risk, impacts the study, or affects completion of the study, in the opinion of the Investigator.
4. Any psychiatric illness that prevents subject from completing the assessments accurately, in the opinion of the Investigator.
5. Subject is a prisoner.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects from all over the United States will be eligible for enrollment as long as they meet the inclusion/exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 211 (Actual)
Dates: Start 2017-06-28 (Actual); Primary Completion 2021-08-03 (Actual); Study Completion 2021-08-03 (Actual)

PRIMARY OUTCOMES:
cervical fusion rate | 12 months
  fusion rate assessed via radiographic confirmation (Xray and CT)

SECONDARY OUTCOMES:
Device Compliance | 6 months
  actual minutes per day device was used compared with prescribed use
revision rate | 12 months
  how many subjects had to be revised at the same level(s) during the course of the study
SF-36 | 12 months
  used to assess the effect of PEMF therapy on the subject's quality of life
Neck Disability Index (NDI) | 12 months
  used to assess the effect of PEMF therapy on the reduction of neck pain
EQ-5D | 12 months
  used to assess the effect of PEMF therapy on quality of life as well as economic impact
VAS pain | 12 months
  used to assess the effect of PEMF therapy on reduction of pain

CONTACTS AND LOCATIONS:
Overall Officials: James T Ryaby, PhD, Principal Investigator — Orthofix Inc.
Locations (1):
- ClinTech Center for Spine Health, Johnstown, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided
if we decide to share, we will share only deidentified summary data